CLINICAL TRIAL: NCT00566527
Title: An Open-label, Randomised, Comparative, Multi-centre Study of the Immunogenicity and Safety of a 2-dose Regimen of ProQuad® Manufactured With rHA Administered to Healthy Children From 9 Months of Age
Brief Title: Comparative Study of Immunogenicity and Safety of a 2-dose Regimen of ProQuad® Manufactured With rHA (V221-038)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V221-038; MRV02C (Other: Sanofi Pasteur Merck Sharp & Dohme (SPMSD) Protocol Number)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: ProQuad® at 9 and 12 months (Experimental): Pediatric participants received ProQuad® Dose 1 at 9 months of age and ProQuad® Dose 2 at 12 months of age.
  Interventions: Biological: ProQuad® manufactured with recombinant Human Albumin (rHA)
- Arm 2: ProQuad® at 11 and 14 months (Experimental): Pediatric participants received ProQuad® Dose 1 at 11 months of age and ProQuad® Dose 2 at 14 months of age.
  Interventions: Biological: ProQuad® manufactured with recombinant Human Albumin (rHA)
- Arm 3: ProQuad at 12 and 15 months (Active Comparator): Pediatric participants received ProQuad® Dose 1 at 12 months of age and ProQuad® Dose 2 at 15 months of age.
  Interventions: Biological: ProQuad® manufactured with recombinant Human Albumin (rHA)

INTERVENTIONS:
Biological: ProQuad® manufactured with recombinant Human Albumin (rHA) — A 2-dose regimen of ProQuad® (0.5 mL per dose) given via subcutaneous injection into the deltoid muscle at a 3-month interval. Each dose contains measles virus Enders' Edmonston strain (live attenuated), mumps virus Jeryl Lynn™ (Level B) strain (live attenuated), rubella virus Wistar RA 27 or 3 strain (live attenuated), and varicella virus Oka or Merck strain (live attenuated).

SUMMARY:
The primary study objectives are:

* To demonstrate that a 2-dose regimen of ProQuad® manufactured with recombinant Human Albumin (rHA) administered at a 3-month interval to healthy children of 11 months of age at the time of Dose 1 is as immunogenic as in healthy children of 12 months of age at the time of Dose 1.
* To demonstrate that a 2-dose regimen of ProQuad® rHA administered at a 3-month interval to healthy children of 9 months of age at the time of Dose 1 is as immunogenic as in healthy children of 12 months of age at the time of Dose 1.
* To demonstrate that a 2-dose regimen of ProQuad® rHA administered at a 3-month interval to healthy children of 11 months of age and 9 months of age at the time of Dose 1 is well-tolerated compared to children of 12 months of age at the time of Dose 1.

The first primary hypothesis was that a 2-dose regimen of ProQuad® rHA, administered at a 3-month interval to children of 11 months of age, would be non-inferior in terms of antibody response rates to measles, mumps, rubella, and varicella at Day 42 following Dose 2, to the same regimen in children of 12 months of age at the time of Dose 1.

If the first primary hypothesis was demonstrated, the second primary hypothesis was that a 2-dose regimen of ProQuad® rHA, administered at a 3-month interval to children of 9 months of age, would be non-inferior in terms of antibody response rates to measles, mumps, rubella, and varicella at Day 42 following Dose 2, to the same regimen in children of 12 months of age at the time of Dose 1.

The secondary study objectives are:

* To describe the antibody titres to measles, mumps, rubella and varicella at Day 42 following Dose 1 and Dose 2 of ProQuad® rHA administered to healthy children from 9 months of age.
* To evaluate the safety profile of Dose 1 and Dose 2 of ProQuad® rHA administered to healthy children from 9 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject of either gender of 9 months of age
2. Negative clinical history of measles, mumps, rubella, varicella or zoster
3. Informed consent form signed by both parents or legal representative
4. Parent(s) or legal representative able to attend all the scheduled visits with the subject and to understand and comply with the study procedures
5. Both parent or legal representative are over 18 years of age
6. Subject is affiliated to a health social security system

Exclusion Criteria:

1. Febrile illness in the previous 3 days
2. Prior vaccination with a measles, mumps, rubella and/or varicella vaccine either alone or in any combination
3. Exposure to measles, mumps, rubella, varicella and/or zoster in the previous 30 days
4. Tuberculin test done in the previous 2 days
5. Severe chronic disease
6. Known active tuberculosis
7. Known personal history of encephalopathy, seizure disorder or progressive, evolving or unstable neurological condition
8. Hereditary problems of fructose intolerance
9. Prior known sensitivity or allergy to any component of the vaccine
10. Known blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems
11. Humoral or cellular immunodeficiency,
12. Immunosuppressive therapy [including systemic corticosteroids (a), given daily or on alternate days at high doses (>=2 mg/kg/day prednisone equivalent or >=20 mg/day if the subject's weight was >10 kg) during at least 14 days in the previous 30 days]
13. Family history of congenital or hereditary immunodeficiency
14. Receipt of immunoglobulins or blood-derived products in the previous 150 days or scheduled to be administered through Visit 5
15. Receipt of an inactivated vaccine in the previous 14 days
16. Receipt of a live non-study vaccine in the previous 28 days
17. Any medical condition which, in the opinion of the investigator, might have interfered with the evaluation of the study objectives
18. Current participation or scheduled participation in any other clinical study through Visit 5

Min Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1620 (Actual)
Dates: Start 2007-11-29 (Actual); Primary Completion 2008-12-29 (Actual); Study Completion 2008-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — SPMSD

REFERENCES:
- [Derived] Vesikari T, Becker T, Gajdos V, Fiquet A, Thomas S, Richard P, Baudin M. Immunogenicity and safety of a two-dose regimen of a combined measles, mumps, rubella and varicella live vaccine (ProQuad((R))) in infants from 9 months of age. Vaccine. 2012 Apr 26;30(20):3082-9. doi: 10.1016/j.vaccine.2012.02.062. Epub 2012 Mar 7. PMID 22406278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric participants from 9 to 12 months of age at the start of the study were recruited at 48 study centers in Finland, France, and Germany.
Groups:
- Arm 1: ProQuad® at 9 and 12 Months: Pediatric participants received ProQuad® Dose 1 at 9 months of age and ProQuad® Dose 2 90 days later at 12 months of age.
- Arm 2: ProQuad® at 11 and 14 Months: Pediatric participants received ProQuad® Dose 1 at 11 months of age and ProQuad® Dose 2 90 days later at 14 months of age.
- Arm 3: ProQuad® at 12 and 15 Months: Pediatric participants received ProQuad® Dose 1 at 12 months of age and ProQuad® Dose 2 90 days later at 15 months of age.
Period: Overall Study
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Started | 541 (Number randomized.) | 540 (Number randomized.) | 539 (Number randomized.)
Received ProQuad® Dose 1 | 529 | 484 | 470
Received ProQuad® Dose 2 | 525 | 478 | 462
Completed | 524 | 474 | 461
Not Completed | 17 | 66 | 78
Not completed — Reason not provided | 3 | 11 | 10
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Physician Decision | 3 | 8 | 20
Not completed — Lost to Follow-up | 3 | 4 | 4
Not completed — Withdrawal by Subject | 6 | 43 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months | Total
Number analyzed (Participants) | 541 | 540 | 539 | 1620
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age at inclusion in study.
  Months | 9.47 (0.29) | 9.48 (0.30) | 9.47 (9.43) | 9.48 (0.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 281 | 258 | 821
  Male | 259 | 259 | 281 | 799

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Arm 2 and Arm 3 Meeting Antibody Immunogenicity Response Criteria Following ProQuad® Dose 2
Description: Immunogenicity response rates were compared in participants with baseline seronegativity from Arm 2 (received ProQuad® Dose 1 at 11 months) and Arm 3 (received ProQuad® Dose 1 at 12 months). Measles, mumps and rubella antibody levels were determined using enzyme-linked immunosorbent assay (ELISA) and varicella antibody levels were determined with glycoprotein-based ELISA (gpELISA). Response and baseline seronegativity criteria were as follows: measles antibody titre ≥255 mIU/mL in participants with baseline titre <255 mIU/mL; mumps antibody titre ≥10 ELISA Ab units/mL in participants with baseline titre <10 ELISA Ab units mL; rubella antibody titre ≥10 IU/mL in participants with baseline titre <10 IU/mL; varicella antibody titre ≥5 gpELISA units/mL in participants with baseline titre <1.25 gpELISA units/mL.
Time Frame: Day 132 (6 weeks after ProQuad® Dose 2)
Population: All baseline seronegative participants with immunogenicity data are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 445 | 443
Percentage of participants
  Measles: number analyzed (Participants) | 440 | 434
  Measles | 98.0 [96.2 to 99.1] | 98.8 [97.3 to 99.6]
  Mumps: number analyzed (Participants) | 436 | 414
  Mumps | 99.5 [98.4 to 99.9] | 99.5 [98.3 to 99.9]
  Rubella | 99.3 [98.0 to 99.9] | 99.5 [98.4 to 99.9]
  Varicella: number analyzed (Participants) | 299 | 347
  Varicella | 100.0 [98.8 to 100.0] | 100.0 [98.9 to 100.0]
Statistical Analysis 1: Comparison: Arm 2: ProQuad® at 11 and 14 Months vs Arm 3: ProQuad® at 12 and 15 Months; Measles difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -5. Values are shown as percentages; Measles Response Rate (Arm 2 - Arm 3) = -0.91, 95% CI 2-sided [-2.82 to 0.87]
Statistical Analysis 2: Comparison: Arm 2: ProQuad® at 11 and 14 Months vs Arm 3: ProQuad® at 12 and 15 Months; Mumps difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -5. Values are shown as percentages; Mumps Response Rate (Arm 2 - Arm 3) = 0.03, 95% CI 2-sided [-1.20 to 1.32]
Statistical Analysis 3: Comparison: Arm 2: ProQuad® at 11 and 14 Months vs Arm 3: ProQuad® at 12 and 15 Months; Rubella difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -5. Values are shown as percentages; Rubella Response Rate (Arm 2 - Arm 3) = -0.22, 95% CI 2-sided [-1.55 to 1.03]
Statistical Analysis 4: Comparison: Arm 2: ProQuad® at 11 and 14 Months vs Arm 3: ProQuad® at 12 and 15 Months; Varicella difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -10. Values are shown as percentages; Varicella Response Rate (Arm 2 - Arm 3) = 0.00, 95% CI 2-sided [-1.28 to 1.10]

2. Primary Outcome: Percentage of Participants in Arm 1 and Arm 3 Meeting Antibody Immunogenicity Response Criteria Following ProQuad® Dose 2
Description: Immunogenicity response rates were compared in participants with baseline seronegativity from Arm 1 (received ProQuad® Dose 1 at 9 months) and Arm 3 (received ProQuad® Dose 1 at 12 months). Measles, mumps and rubella antibody levels were determined using ELISA and varicella antibody levels were determined with gpELISA. Response and baseline seronegativity criteria were as follows: measles antibody titre ≥255 mIU/mL in participants with baseline titre <255 mIU/mL; mumps antibody titre ≥10 ELISA Ab units/mL in participants with baseline titre <10 ELISA Ab units mL; rubella antibody titre ≥10 IU/mL in participants with baseline titre <10 IU/mL; varicella antibody titre ≥5 gpELISA units/mL in participants with baseline titre <1.25 gpELISA units/mL.
Time Frame: Day 132 (6 weeks after ProQuad® Dose 2)
Population: All baseline seronegative participants with immunogenicity data are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 500 | 443
Percentage of participants
  Measles: number analyzed (Participants) | 490 | 434
  Measles | 94.9 [92.6 to 96.7] | 98.8 [97.3 to 99.6]
  Mumps: number analyzed (Participants) | 484 | 414
  Mumps | 99.2 [97.9 to 99.8] | 99.5 [98.3 to 99.9]
  Rubella | 99.4 [98.3 to 99.9] | 99.5 [98.4 to 99.9]
  Varicella: number analyzed (Participants) | 208 | 347
  Varicella | 100.0 [98.2 to 100.0] | 100.0 [98.9 to 100.0]
Statistical Analysis 1: Comparison: Arm 1: ProQuad® at 9 and 12 Months vs Arm 3: ProQuad® at 12 and 15 Months; Measles difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -5. Values are shown as percentages; Measles Response Rate (Arm 1 - Arm 3) = -3.97, 95% CI 2-sided [-6.44 to -1.87]
Statistical Analysis 2: Comparison: Arm 1: ProQuad® at 9 and 12 Months vs Arm 3: ProQuad® at 12 and 15 Months; Mumps difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -5. Values are shown as percentages; Mumps Response Rate (Arm 1 - Arm 3) = -0.35, 95% CI 2-sided [-1.71 to 1.01]
Statistical Analysis 3: Comparison: Arm 1: ProQuad® at 9 and 12 Months vs Arm 3: ProQuad® at 12 and 15 Months; Rubella difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -5. Values are shown as percentages; Rubella Response Rate (Arm 1 - Arm 3) = -0.15, 95% CI 2-sided [-1.34 to 1.09]
Statistical Analysis 4: Comparison: Arm 1: ProQuad® at 9 and 12 Months vs Arm 3: ProQuad® at 12 and 15 Months; Varicella difference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared when the lower bound of the 95% CI was > -10. Values are shown as percentages; Varicella Response Rate (Arm 1 - Arm 3) = 0.00, 95% CI 2-sided [-1.83 to 1.10]

3. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Reactions
Description: The solicited injection-site AEs erythema, swelling, and pain were monitored for 4 days after administration of ProQuad® Dose 1.
Time Frame: Day 1 to Day 4 (up to 4 days after ProQuad® Dose 1)
Population: All participants who received ProQuad® Dose 1 and have safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 528 | 480 | 466
Percentage of participants
  Injection-site erythema | 14.4 [11.5 to 17.7] | 15.4 [12.3 to 19.0] | 17.2 [13.9 to 20.9]
  Injection-site pain | 11.4 [8.8 to 14.4] | 10.4 [7.8 to 13.5] | 13.7 [10.7 to 17.2]
  Injection-site swelling | 2.3 [1.2 to 3.9] | 4.6 [2.9 to 6.9] | 2.4 [1.2 to 4.2]

4. Primary Outcome: Percentage of Participants Experiencing Unsolicited Injection-site Adverse Reactions
Description: The percentage of participants with unsolicited injection-site reactions after ProQuad® Dose 1 was determined.
Time Frame: Up to Day 28 (up to 28 days after ProQuad® Dose 1)
Population: All participants who received ProQuad® Dose 1 and have safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 528 | 480 | 466
Percentage of participants | 24.8 [21.2 to 28.7] | 23.3 [19.6 to 27.4] | 19.1 [15.6 to 23.0]

5. Primary Outcome: Percentage of Participants Experiencing a Systemic Adverse Event After ProQuad® Dose 1
Description: The percentage of participants with systemic adverse events after ProQuad® Dose 1 was determined.
Time Frame: Up to Day 28 (up to 28 days after ProQuad® Dose 1)
Population: All participants who received ProQuad® Dose 1 and have safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 528 | 480 | 466
Percentage of participants | 72.0 [67.9 to 75.8] | 71.9 [67.6 to 75.9] | 71.9 [67.6 to 75.9]

6. Primary Outcome: Percentage of Participants With Rectal (or Rectal Equivalent) Temperature ≥ 39.4°C
Description: The percentage of participants with a rectal (or rectal equivalent) temperature ≥ 39.4°C after ProQuad® Dose 1 was determined.
Time Frame: Up to Day 28 (up to 28 days after ProQuad® Dose 1)
Population: All participants who received ProQuad® Dose 1 and have safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 528 | 480 | 466
Percentage of participants | 8.8 [6.5 to 11.5] | 10.3 [7.7 to 13.4] | 14.8 [11.7 to 18.4]

7. Secondary Outcome: Geometric Mean Titres (GMT) to Measles, Mumps, Rubella, and Varicella After ProQuad® Dose 1
Description: Antibody titres (GMT) to measles, mumps, rubella, and varicella were determined after the first ProQuad® dose in participants with seronegative baseline values. Baseline seronegativity criteria were as follows: measles antibody titre <255 mIU/mL; mumps antibody titre <10 ELISA Ab units mL; rubella antibody titre <10 IU/mL; and varicella antibody titre <1.25 gpELISA units/mL.
Time Frame: Day 42 (6 weeks after ProQuad® Dose 1)
Population: All participants with seronegative baselines who received ProQuad® Dose 1 and have immunogenicity data available are included.
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 518 | 460 | 447
GMT
  Measles (mIU/mL): number analyzed (Participants) | 508 | 455 | 438
  Measles (mIU/mL) | 942 [808 to 1098] | 1977 [1736 to 2252] | 2500 [2199 to 2841]
  Mumps (ELISA Ab units/mL): number analyzed (Participants) | 499 | 453 | 417
  Mumps (ELISA Ab units/mL) | 73 [68 to 79] | 91 [84 to 99] | 86 [79 to 93]
  Rubella (IU/mL) | 64 [60 to 70] | 77 [71 to 83] | 81 [75 to 88]
  Varicella (gpELISA units/mL): number analyzed (Participants) | 220 | 312 | 353
  Varicella (gpELISA units/mL) | 15 [13 to 16] | 15 [14 to 16] | 15 [14 to 16]

8. Secondary Outcome: GMT to Measles, Mumps, Rubella, and Varicella After ProQuad® Dose 2
Description: Antibody titres (GMT) to measles, mumps, rubella, and varicella were determined after the second ProQuad® dose in participants with seronegative baseline values. Baseline seronegativity criteria were as follows: measles antibody titre <255 mIU/mL; mumps antibody titre <10 ELISA Ab units mL; rubella antibody titre <10 IU/mL; and varicella antibody titre <1.25 gpELISA units/mL.
Time Frame: Day 132 (6 weeks after ProQuad® Dose 2)
Population: All participants with seronegative baselines who received ProQuad® Dose 2 and have immunogenicity data available are included.
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 500 | 445 | 443
GMT
  Measles (mIU/mL): number analyzed (Participants) | 490 | 440 | 434
  Measles (mIU/mL) | 1817 [1645 to 2006] | 2320 [2129 to 2529] | 2703 [2492 to 2933]
  Mumps (ELISA Ab units/mL): number analyzed (Participants) | 481 | 436 | 414
  Mumps (ELISA Ab units/mL) | 157 [147 to 168] | 163 [151 to 175] | 172 [159 to 185]
  Rubella (IU/mL) | 106 [99 to 113] | 116 [109 to 124] | 118 [111 to 126]
  Varicella {gpELISA units/mL): number analyzed (Participants) | 208 | 299 | 347
  Varicella {gpELISA units/mL) | 431 [372 to 500] | 460 [410 to 517] | 515 [466 to 569]

9. Secondary Outcome: Percentage of Participants With Varicella Antibody Titre ≥ 1.25 gpELISA Units/mL
Description: The percentage of participants with varicella antibody titre ≥ 1.25 gpELISA units/mL 6 weeks after each ProQuad® dose was determined.
Time Frame: Day 132 (6 weeks after ProQuad® Dose 2)
Population: All participants who received ProQuad® and have serology results are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 523 | 474 | 459
Percentage of participants
  ProQuad® Dose 1: number analyzed (Participants) | 523 | 474 | 458
  ProQuad® Dose 1 | 99.8 [98.9 to 100.0] | 100.0 [99.2 to 100.0] | 99.8 [98.8 to 100.0]
  ProQuad® Dose 2: number analyzed (Participants) | 521 | 469 | 459
  ProQuad® Dose 2 | 100.0 [99.3 to 100.0] | 100.0 [99.2 to 100.0] | 100.0 [99.2 to 100.0]

10. Secondary Outcome: Percentage of Baseline Seronegative Participants Meeting Antibody Immunogenicity Response Criteria After ProQuad® Dose 1
Description: The percentage of baseline seronegative participants meeting measles, mumps, rubella, and varicella antibody response criteria after the first ProQuad® dose was determined. Measles, mumps and rubella antibody levels were determined using ELISA and varicella antibody levels were determined with gpELISA. Response and baseline seronegativity criteria were as follows: measles antibody titre ≥255 mIU/mL in participants with baseline titre <255 mIU/mL; mumps antibody titre ≥10 ELISA Ab units/mL in participants with baseline titre <10 ELISA Ab units mL; rubella antibody titre ≥10 IU/mL in participants with baseline titre <10 IU/mL; varicella antibody titre ≥5 gpELISA units/mL in participants with baseline titre <1.25 gpELISA units/mL.
Time Frame: Day 42 (6 weeks after ProQuad® Dose 1)
Population: All baseline seronegative participants with immunogenicity data are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 518 | 460 | 447
Percentage of participants
  Measles: number analyzed (Participants) | 508 | 455 | 438
  Measles | 72.6 [68.5 to 76.5] | 87.9 [84.6 to 90.8] | 90.2 [87.0 to 92.8]
  Mumps: number analyzed (Participants) | 499 | 453 | 417
  Mumps | 96.6 [94.6 to 98.0] | 98.7 [97.1 to 99.5] | 98.3 [96.6 to 99.3]
  Rubella | 97.7 [96.0 to 98.8] | 98.9 [97.5 to 99.6] | 98.0 [96.2 to 99.1]
  Varicella: number analyzed (Participants) | 220 | 312 | 353
  Varicella | 95.0 [91.2 to 97.5] | 97.8 [95.4 to 99.1] | 97.5 [95.2 to 98.8]

11. Secondary Outcome: Percentage of Participants With Non-injection Site Rashes of Interest Following ProQuad® Dose 1
Description: The percentage of participants with rashes of interest after ProQuad® Dose 1 was determined. Rashes of interest consisted of measles-like rash, rubella-like rash, varicella-like rash, zoster-like rash, and mumps-like rash.
Time Frame: Up to Day 28 (up to 4 weeks after ProQuad® Dose 1)
Population: All participants who received ProQuad® Dose 1 and have safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 528 | 480 | 466
Percentage of participants
  Measles-like rash | 4.0 [2.5 to 6.0] | 5.8 [3.9 to 8.3] | 6.9 [4.7 to 9.6]
  Rubella-like rash | 1.3 [0.5 to 2.7] | 1.9 [0.9 to 3.5] | 1.5 [0.6 to 3.1]
  Varicella-like rash | 5.3 [3.6 to 7.6] | 4.0 [2.4 to 6.1] | 6.4 [4.4 to 9.1]
  Zoster-like rash | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Mumps-like illness | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.4 [0.1 to 1.5]

12. Secondary Outcome: Percentage of Participants With Non-injection Site Rashes of Interest Following ProQuad® Dose 2
Description: The percentage of participants with rashes of interest after receiving ProQuad® Dose 2 was determined. Rashes of interest consisted of measles-like rash, rubella-like rash, varicella-like rash, zoster-like rash, and mumps-like rash.
Time Frame: Day 132 (6 weeks after ProQuad® Dose 2)
Population: All participants who received ProQuad® Dose 2 and have safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Number analyzed (Participants) | 524 | 474 | 462
Percentage of participants
  Measles-like rash | 2.1 [1.1 to 3.7] | 2.7 [1.5 to 4.6] | 2.8 [1.5 to 4.8]
  Rubella-like rash | 1.5 [0.7 to 3.0] | 1.9 [0.9 to 3.6] | 0.9 [0.2 to 2.2]
  Varicella-like rash | 2.1 [1.1 to 3.7] | 3.8 [2.3 to 5.9] | 2.6 [1.3 to 4.5]
  Zoster-like rash | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Mumps-like illness | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Up to 146 days (up to 56 days after Dose 2)
Description: An adverse event is any untoward medical occurrence in a participant administered an investigational medicinal product (IMP) and which does not necessarily have a causal relationship with the IMP. Participants who received at least one dose of ProQuad® and have follow-up data available are included.
Arm/Group | Arm 1: ProQuad® at 9 and 12 Months | Arm 2: ProQuad® at 11 and 14 Months | Arm 3: ProQuad® at 12 and 15 Months
Serious Adverse Events (participants affected / at risk) | 21/541 | 15/540 | 17/539
Other Adverse Events (participants affected / at risk) | 468/541 | 430/540 | 401/539
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: ProQuad® at 9 and 12 Months (N=541) | Arm 2: ProQuad® at 11 and 14 Months (N=540) | Arm 3: ProQuad® at 12 and 15 Months (N=539)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 4 (5) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Gastroenteritis Norwalk virus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 6 (6) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (4)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: ProQuad® at 9 and 12 Months (N=541) | Arm 2: ProQuad® at 11 and 14 Months (N=540) | Arm 3: ProQuad® at 12 and 15 Months (N=539)
Diarrhoea (Gastrointestinal disorders) | 66 (71) | 62 (77) | 62 (72)
Teething (Gastrointestinal disorders) | 44 (65) | 28 (39) | 26 (32)
Vomiting (Gastrointestinal disorders) | 37 (44) | 26 (31) | 23 (28)
Injection site erythema (General disorders) | 278 (383) | 262 (350) | 233 (322)
Injection site pain (General disorders) | 99 (126) | 100 (123) | 109 (137)
Injection site swelling (General disorders) | 107 (117) | 90 (100) | 82 (92)
Irritability (General disorders) | 77 (127) | 70 (103) | 86 (113)
Pyrexia (General disorders) | 92 (117) | 92 (133) | 76 (99)
Ear infection (Infections and infestations) | 40 (44) | 24 (28) | 27 (31)
Gastroenteritis (Infections and infestations) | 28 (29) | 30 (30) | 15 (16)
Nasopharyngitis (Infections and infestations) | 51 (58) | 42 (51) | 37 (42)
Otitis media (Infections and infestations) | 45 (53) | 46 (50) | 41 (48)
Rhinitis (Infections and infestations) | 101 (127) | 94 (110) | 75 (99)
Upper respiratory tract infection (Infections and infestations) | 70 (85) | 68 (87) | 76 (98)
Crying (Psychiatric disorders) | 36 (43) | 17 (29) | 19 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 61 (68) | 45 (52) | 40 (44)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 34 (38) | 26 (28) | 30 (40)
Rash (Skin and subcutaneous tissue disorders) | 52 (64) | 37 (47) | 41 (48)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 32 (33) | 39 (41) | 41 (45)
Rash vesicular (Skin and subcutaneous tissue disorders) | 35 (39) | 34 (40) | 39 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sanofi Pasteur MSD shall have sixty days to review these documents and may refuse to give its consent in part or whole for confidential reasons (including but not limited to intellectual property rights, whether patentable or not).